CLINICAL TRIAL: NCT05589922
Title: Determining the Relationship Between Abnormal Modified Schober Index and Demographic Characteristics and Clinical Variables in Patients With Ankylosing Spondylitis
Brief Title: The Relationship Between Abnormal Modified Schober Index and Demographic Characteristics and Clinical Variables
Status: Completed | Type: Observational
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Gamze Kus, assistant professor, Mustafa Kemal University
Other Study IDs: MustafaKU07
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Spinal mobility; Kinesiophobia; Balance
MeSH Terms: conditions — Spondylitis, Ankylosing; Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with abnormal modified Schober index: This group will include the patients with Ankylosing Spondylitis who have modified Schober index smaller than 5 cm
- Patients with normal modified Schober index: This group will include the patients with Ankylosing Spondylitis who have modified Schober index bigger than 5 cm

SUMMARY:
This study will aim to compare ankylosing spondylitis (AS) participants with abnormal modified Schober index (AMSI) versus AS participants with normal modified Schober index (NMSI) in pain, morning stiffness, balance, kinesiophobia and the fear of falling. In addition, the investigators will aim to determine which demographic characteristics and variables predispose AMSI to occur

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS), a common type of spondyloarthropathy, is a chronic inflammatory disease that affects spinal joints, and adjacent soft tissues such as sacroiliac joints, tendons, and entheses (1). Inflammation of the spinal structures and progressive changes in the surrounding tissue is largely responsible for decreased physical function and mobility in participants with AS (2).

It is unknown how these parameters of AS participants with AMSI (smaller than 5 cm) are affected compared to AS participants with normal modified Schober index (NMSI, bigger than 5 cm). In addition, it is unclear which demographic characteristics and variables predispose AMSI to occur.

This study will aim to compare AS participants with abnormal modified Schober index (AMSI) versus AS participants with normal modified Schober index (NMSI) in pain, morning stiffness, balance, kinesiophobia and the fear of falling. In addition, the investigators will aim to determine which demographic characteristics and variables predispose AMSI to occur

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet the modified New York criteria for AS
* Participants over 18 years

Exclusion Criteria:

* Participants with other concomitant rheumatic diseases (such as fibromyalgia, rheumatoid arthritis, etc.),
* Participants with cognitive or psychiatric disorders,
* Participants with neuromuscular or orthopedic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ankylosing Spondylitis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Modified Schober Index | at baseline
  The measurement of the MSI starts with the subject in an upright posture. After being determined the posterior superior iliac spines, a horizontal line is drawn at the center of both posterior superior iliac spines. Ten cm above and five cm below the first line are marked. The distance between the top and bottom line is remeasured after the patient attempts to flex forward as far as possible while keeping the knees straight
Bath AS Metrology Index (BASMI) | at baseline
  The BASMI is evulated quantify the mobility of the axial skeleton and includes assessments of lateral lumbar flexion, tragus-to-wall distance, lumbar flexion, intermalleolar distance, and cervical rotation. Each measure is assigned a score of 0 to 2 with the higher score indicating greater impairment in mobility
Timed up and go test | at baseline
  It aims to assess mobility and balance. It measures the time in seconds for a subject to stand up from an armchair, walk 3 m, turn, walk back to the chair, and sit down
tandem stance test | At baseline
  For the tandem stance test, patients stand holding onto a railing while placing one foot in front of the other. The researcher standing behind the patient starts timing when the patient's contact with the railing is released. It is recorded for 30 seconds or until participants contact external support or move out of tandem stance
Falls Efficacy Scale-International | At baseline
  The FES-I consists of 16 questions questioning how confident patients are in performing activities without falling. According to the answers, each question is scored between 1 and 4 (1 = not at all concerned, 4 = very concerned), and a higher score is associated with a greater fear of falling
Tampa Scale for Kinesiophobia | At baseline
  The TSK contains 17 questions which measures fear of movement and/or reinjury. The scale uses 4-point Likert scoring (1 = entirely disagree, 4 = entirely agree). A total score ranges from 11 to 44 points and a cut-off point was determined as ≥37 points indicate a high kinesiophobia level

SECONDARY OUTCOMES:
functional reach test | At baseline
  For the functional reach test, the patient is asked to stand erect with feet separated from each other in a comfortable position and reach the farthest distance without touching the wall or without taking a step. The difference in the distance between the starting point and the endpoint is recorded in cm.
30-second chair sit-to-stand test | At baseline
  The proximal muscle strength and endurance of the lower extremities assessed by the 30-second chair sit-to-stand. The patients is seated in an armless chair with their back straight, arms crossed in front of the chest, and feet approximately a shoulder width apart and placed on the floor. Then patients are instructed to fully sit between each stand.
single leg stance test | At baseline
  For the SLST is performed by standing on one leg (eyes open) barefoot for 20 seconds, the other knee flexed without touching the other leg, with arms are crossed. The test will be repeated thrice on each foot, and the average time will be used for analysis.
finger-to-floor distance measure | At baseline
  For finger-to-floor distance (FFD), the subject is asked to perform maximal lumbar flexion while keeping the knees extend. After which, the distance between the right middle finger and the floor is measured using a tape measure
Visual Analogue Scale | At baseline
  Pain scores of the patients at night, at rest, and during activity are measured using visual analogue scale (VAS). (0-10 mm; 0 indicates no pain and 10 indicates severe pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University, Faculty of Health Science, Department of Physiotherapy and Rehabilitation, Hatay, Alahan, Turkey (Türkiye)